CLINICAL TRIAL: NCT06528561
Title: Impact of a Physical Exercise Program on the Self-care Capacity of People Hospitalized for Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar Universitário de Santo António (Other)
Responsible Party: Principal Investigator, Ivo Lopes, Specialist Nurse, Centro Hospitalar Universitário de Santo António
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.226(186-DEFI/178-CE)
Record Dates: First submitted 2024-07-20; First posted 2024-07-30 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure
Keywords: self-care; heart failure; rehabilitation nursing; exercise
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Self-care program
  Interventions: Procedure: Sef-care program with exercise
- Control group (Active Comparator): EarlyRehabilitation in Cardiology-Heart Failure program (ERIC-HF)
  Reference: Delgado B, Lopes I, Gomes B, Novo A. Early rehabilitation in cardiology - heart failure: The ERIC-HF protocol, a novel intervention to decompensated heart failure patients rehabilitation. Eur J Cardiovasc Nurs. 2020 Oct;19(7):592-599. doi: 10.1177/1474515120913806. Epub 2020 Apr 22.
  Interventions: Procedure: Sef-care program with exercise

INTERVENTIONS:
Procedure: Sef-care program with exercise — Self-care program with physical exercise with aerobic and muscular strength components implemented progressively according to the participant's clinical evolution

SUMMARY:
The objective of the study is to evaluate the effectiveness of a self-care program that integrates physical exercise with components of aerobic and muscular strength training in improving functional capacity and muscular strength in people hospitalized for decompensated heart failure, in a clinical stabilization phase

The main question it aims to answer is:

Is the Self-care program that integrates physical exercise with aerobic and muscular strength training components effective in improving the capacity for self-care in people hospitalized for decompensated HF, in the clinical stabilization phase?

In this randomized clinical trial, the Self-Care program will be applied in the experimental group. The ERIC-HF program will be applied in the control group. The ERIC-HF is a program of exercise only with an aerobic component.

Participants will complete these programs during their hospital stay and various assessment instruments (quality of life, functional capacity, capacity for self-care, muscle strength) will be applied at admission, at discharge and one month after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Participants: Clinical diagnosis of decompensated HF, regardless of etiology or ventricular function;
* Participants: Be over 18 years old;
* Participants: Be able to provide informed consent.

Exclusion Criteria (participants):

* Osteoarticular pathology that causes physical limitations that prevent the performance of physical exercise;
* Existence of intravenous inotropic medication;
* Uncontrolled auricular or ventricular arrhythmias;
* Chest pain in the last 8 hours;
* Heart rate greater than 120;
* Dyspnea at rest;
* Uncontrolled blood pressure - Systolic blood pressure greater than 180mmHg or diastolic blood pressure greater than 110mmHg;
* 2nd or 3rd degree atrioventricular block;
* Oxygen need at a rate greater than 3L/min;
* Glycemic decompensation in the last 12 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
functional capacity - distance covered in meters with the use of the 6 Minute Walk Test | immediately after the intervention (at discharge from hospitalization)
  The 6MWT is one of the most widely used instruments to assess an individual's tolerance to exertion. It reflects functional capacity, participant gait autonomy, and effectiveness of the physical exercise training This test should be performed in a 30 to 50 meter corridor that is familiar to the individual. The person is asked to walk as fast as possible over a period of six minutes.
Hand Grip Strength Test | baseline, pre-intervention (upon admission) and immediately after the intervention (at discharge from hospitalization)
  Hand grip strength is essential for performing various daily activities, being a predictive factor of functional capacity, all-cause mortality, cardiac mortality, and predictive of hospital readmission due to decompensated heart failure. It is a force assessment test that measures force production in kilograms. It is easy to apply, and the participant must perform 3 measurements with a dynamometer and the average value calculated is accepted.
Self-care skills assessed using the Self-Care of Heart Failure Index | baseline, pre-intervention (upon admission) and one month after the intervention and discharge from hospitalization
  This instrument allows the assessment of self-care in the maintenance, management and self-confidence stages of people with heart failure, allowing the identification of the stage(s) in which self-care is compromised. The scale consists of twenty-two items, distributed in three subscales called sections A, B and C. Section A consists of 10 items and is related to the maintenance of self-care. Section B consists of six items related to self-care management. Section C is composed of six items related to confidence in self-care.

SECONDARY OUTCOMES:
Impact of dyspnea on the various activities of daily living, assessed using the London Chest Activity of Daily Living | baseline, pre-intervention (upon admission) and immediately after the intervention (at discharge from hospitalization)
  This scale evaluates the impact of dyspnea on the various activities of daily living (ADL), in order to measure its limitation. This questionnaire consists of 15 items that are divided into four domains related to personal care, domestic activities, physical activities and leisure, allowing the assessment of the person's degree of dyspnea and the response to a therapeutic intervention. Each of the items is assigned a score from 0 to 5, in which higher values indicate greater limitation in ADL due to dyspnea. A partial score can be obtained for each domain or a global assessment of the scale with a maximum score of 75 points can be used. Given that the program is applied in the context of hospitalization, the partial score is chosen, and the components related to domestic care are not evaluated, and thus the maximum score to be obtained will be 45.
Functional performance of the lower limbs assessed through the score obtained using the Short physical performance battery | baseline, pre-intervention (upon admission) and immediately after the intervention (at discharge from hospitalization)
  This instrument consists of 3 components - orthostatic balance test in 3 different positions, test of the gait speed that the participant can achieve in a 4-meter course and test evaluation of the time it takes the participant to perform 5 repetitions of getting up and sitting down from a chair. The total score varies between 0 and 12 points, in which the highest value corresponds to better mobility and muscle strength of the lower limbs. It is an instrument that is easy to apply and can be used in an inpatient context. A final score lower than 10 is predictive of mortality and hospital readmission. This instrument is valid for inferring about the function and muscle strength of people's lower limbs, which is very useful in the heart failure population, in which loss of muscle mass and strength are generally present and affect tolerance to exertion and competence in the execution of ADLs.
Quality of life perceived assessed using The Minnesota Living with Heart Failure Questionnaire | baseline, pre-intervention (upon admission) and one month after the intervention and discharge from hospitalization
  This self-completion tool consists of 21 questions that address the impact of heart failure on physical, emotional and social levels, and the person can choose an answer option ranging from 0 (not applicable), 1 (very little) to 5 (too much). Thus, the total score can vary between 0 and 105, and the greater the sum of the results of all the questions, the greater the impact of the heart failure on the person's life. This scale is also used to assess whether a particular treatment or clinical program for heart failure improves the quality of life of individuals by reducing the adverse effects that the disease causes.

CONTACTS AND LOCATIONS:
Overall Officials: Ivo Lopes, Principal Investigator — Centro Hospitalar Universitário de Santo António
Locations (1):
- Centro Hospitalar Universitário de Santo António - ULS Santo António, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR